CLINICAL TRIAL: NCT02732106
Title: Characterization of Adipose Derived Regenerative Cells (ADRCs) From Excess Tissue and Cells Designated for Discard From Patients With Chronic Heart Disease
Brief Title: Characterization of Adipose Derived Regenerative Cells (ADRCs) From Patients With Chronic Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: CYTX-01
Record Dates: First submitted 2014-11-19; First posted 2016-04-08 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Heart Failure
Keywords: ADRCs, cell characterization

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Human adipose tissue is now recognized as an acceptable, highly abundant source of adipose-derived regenerative cells (ADRCs). ADRCs are a heterogeneous or mixed population of cells found in adipose tissue including adult stem cells, leukocytes, connective tissue and vessel-associated cells. Autologous adult regenerative cells are thought to promote healing of scarred or injured tissue. While the investigators are learning more about the exact mechanisms every day, it is believed that this heterogeneous population of cells influences the local environment via cell-to-cell signaling, immune modulation, and differentiation into other cell types. The use of ADRCs in the treatment of many different medical conditions (including cardiovascular disease, soft tissue defects, wound healing, and many more) is being evaluated in numerous clinical and preclinical studies around the world. While there is a considerable amount of information regarding the cellular composition of ADRCs isolated from healthy donors, basically there is no much data regarding the ADRC composition from cardiac patients. In this study, adipose tissue or cells from chronic heart ischemia patients, that would otherwise be thrown away in waste, will be provided to researchers who will study these cells with the objective to characterize ADRCs derived from patients with a heart disease and to compare if a heart disease state does impact ADRC cell composition.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the ATHENA clinical trial that donated their leftover material to be studied.

Exclusion Criteria:

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic heart disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Adipose-Derived Regenerative Cells (ADRCs)- Cell Characterization | Day 1
  Cells will be evaluated regarding cell composition by flow cytometric assays.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kesten, MD, Principal Investigator — Cytori Therapeutics
Locations (4):
- United States (4):
  - Scripps Clinic - Torrey Pines, Scripps Green Hospital, La Jolla, California
  - University of Florida, Gainesville, Florida
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Texas Heart Institute, Houston, Texas